CLINICAL TRIAL: NCT01636336
Title: Effects of Progesterone on Smoked Nicotine Induced Changes in Hormones and Subjective Ratings of Stimulant Drug Effects
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical studies are stopped, pending funding
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Nancy Kishlar Mello, Director, Alcohol and Drug Abuse Research Center & Professor of Psychology (Neuroscience), Harvard Medical School, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2009-p-001665
Record Dates: First submitted 2012-06-21; First posted 2012-07-10 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Progesterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Female Smokers (Mid-Luteal Phase; cycle days 18-22) (Active Comparator)
  Interventions: Other: Nicotine; Other: Progesterone
- Female Smokers (Early Follicular Phase; cycle days 4-8) (Active Comparator)
  Interventions: Other: Nicotine; Other: Progesterone

INTERVENTIONS:
Other: Nicotine — Two doses of nicotine will be utilized in the study: a commercially available, high-yield nicotine cigarette (Marlboro Red; Phillip Morris brand) and a denicotinized cigarette (Murty Pharmaceuticals Inc., Lexington, KY). The high dose cigarettes contain 15.48 mg of nicotine and 16 mg of tar based on analysis by the Massachusetts Department of Public Health (MDPH, 1998). The low nicotine cigarettes contain 1.1 mg of nicotine and deliver 0.1 mg of nicotine and 2.8 mg of tar based on analyses provided by the manufacturer.
Other: Progesterone — Prometrium capsules containing 200 mg of micronized progesterone will be obtained from Solvay Pharmaceuticals, Inc. (210 Main Street West, Baudette, MN, 56623, phone (218) 634-3500, fax (218) 634-3540).

SUMMARY:
The clinical studies propose to study the abuse-related effects of nicotine after progesterone administration during the follicular phase in women of reproductive age. Concurrent analysis of hypothalamic-pituitary-adrenal hormones should help to clarify the role of the HPA axis in the abuse-related effects of nicotine.

DETAILED DESCRIPTION:
These clinical studies will analyze the interactions between progesterone, nicotine, alterations in endocrine hormones, mood and cardiovascular measures. The studies also intend to examine the contribution of menstrual cycle phase. It is hypothesized that this novel focus on nicotine's rapid hormonal, cardiovascular and subjective effects will be important for developing novel biologic approaches to treatment for nicotine abuse and dependence as well as advancing our understanding of the neurobiology of nicotine reinforcement.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 40 who currently smoke at least 15 cigarettes every day, and who fulfill DSM-IV diagnostic criteria for nicotine dependence will be eligible for participation.
* No evidence of clinically significant disease based upon complete medical history and physical examination supervised by Dr. Arthur Siegel (Chief of Internal Medicine).
* Absence of DSM-IV Axis I Disorders other than nicotine dependence (305.10) as measured by the Structured Clinical Interview (SCID).
* Routine laboratory blood tests including complete blood count, electrolytes, BUN and creatinine, liver function tests, hepatitis panel and urinalysis will be performed. Laboratory parameters must be within the normal range. HBsAg must be negative but subjects who have hepatitis serology consistent with previous exposure to Hepatitis A, Hepatitis B, or Hepatitis C, but who do not have clinical and biochemical evidence of acute infection, will be acceptable.
* Hematocrit levels ≥ 35% for females.
* Serum pregnancy test (hCG beta subunit) results must be negative within 24 hrs of the study session day.
* Normal EKG.
* A Body Mass Index (BMI-ratio of weight (W) to height (H) squared; W/H2=kg/m2) of between 18.0 and 27.0 for women.
* Subjects must be able to read and understand instructions, as well as provide a valid informed consent.

Exclusion Criteria:

* Participants with any lifetime DSM-IV Axis I disorder other than nicotine dependence.
* Participants with clinically significant medical disorders.
* Women who are pregnant as determined by laboratory testing for serum beta hCG.
* Women who use hormonal contraceptive medications will not be accepted, because this would confound the hormonal measures.
* Women with a mean BMI of outside the range 18.0-27.0.
* Participants who describe themselves as seeking treatment will not be selected but will be referred to local smoking cessation programs.
* Subjects with peanut/peanut oil allergies will be excluded.
* Participants diagnosed with lactose intolerance will be excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Effects of Progesterone on Nicotine-Induced Changes on the hypothalamic-pituitary adrenal (HPA) axis | From baseline to study completion (approximately 8 months for females)
  The investigators are examining the effects of progesterone on smoked nicotine induced changes in serum/plasma hormone levels.
Effects of Nicotine on the hypothalamic-pituitary-gonadal (HPG) axis | From baseline to study completion (approximately 8 months for females)
  The investigators are examining the effects of smoked nicotine on serum nicotine levels and serum/plasma hormone levels.

SECONDARY OUTCOMES:
Effects of Nicotine on a Visual Analog Scale of Mood States | From baseline to study completion (approximately 8 months for females)
  The investigators are examining the effects of progesterone on smoked nicotine induced changes in subjective states ("high," "like," "rush," "dizzy," etc.), as measured by a visual analog scale.
Effects of Nicotine on Cardiovascular Measures | From baseline to study completion (approximately 8 months for females)
  The investigators are examining the effects of progesterone on smoked nicotine induced changes in cardiovascular measures, as measured by blood pressure and heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Mello, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- Alcohol and Drug Abuse Research Center at McLean Hospital, Belmont, Massachusetts, United States